CLINICAL TRIAL: NCT01413776
Title: Effects of a Fortified Dietary Supplement for Pregnant Women on Maternal and Newborn Outcomes in Kampong Chhnang Province, Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: International Relief and Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H11-00801
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Maternal and Newborn Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement (Experimental): Pregnant women in 37 villages.
  Interventions: Dietary Supplement: Corn Soya Blend+
- Control group (No Intervention): Pregnant women in 38 villages

INTERVENTIONS:
Dietary Supplement: Corn Soya Blend+ — A blended food consisting of corn (75-80%) and soybeans (20-25%) that has been fortified with a premix of 19 vitamins and minerals.
  Arms: Dietary supplement

SUMMARY:
The study will evaluate the effects of a nutrition supplement for pregnant women on birth weight and other outcomes. The hypothesis is pregnant women who consume a daily fortified food supplement will produce babies with a higher mean birth weight than those who do not.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* in first trimester of pregnancy
* plans to reside in the same village during the entire pregnancy

Exclusion Criteria:

* a minor
* not in first trimester of pregnancy
* plans to relocate during the pregnancy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 547 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mean birth weight | 9 months

SECONDARY OUTCOMES:
Mean gestational weight gain | 9 months
Mean maternal hemoglobin level | 9 months
Mean birth length and head circumference | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Judy McLean, Dr., Principal Investigator — University of British Columbia
Locations (1):
- 4 Health Centers, Kampong Chhnang, Cambodia

REFERENCES:
- [Derived] Janmohamed A, Karakochuk CD, Boungnasiri S, Chapman GE, Janssen PA, Brant R, Green TJ, McLean J. Prenatal supplementation with Corn Soya Blend Plus reduces the risk of maternal anemia in late gestation and lowers the rate of preterm birth but does not significantly improve maternal weight gain and birth anthropometric measurements in rural Cambodian women: a randomized trial. Am J Clin Nutr. 2016 Feb;103(2):559-66. doi: 10.3945/ajcn.114.104034. Epub 2016 Jan 6. PMID 26739037
- [Derived] Janmohamed A, Karakochuk CD, Boungnasiri S, Whitfield KC, Chapman GE, Janssen P, McLean J, Green TJ. Factors affecting the acceptability and consumption of Corn Soya Blend Plus as a prenatal dietary supplement among pregnant women in rural Cambodia. Public Health Nutr. 2016 Jul;19(10):1842-51. doi: 10.1017/S1368980015003018. Epub 2015 Oct 16. PMID 26471409